CLINICAL TRIAL: NCT00772226
Title: The Use of Music as Pain Therapy in Patients Undergoing Laparoscopic Cholecystectomy in a Day Care Unit
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Randers Regional Hospital (Other)
Responsible Party: Principal Investigator, Thorbjorn Sommer, Consultant M.D, Ph.D ass Proff, Randers Regional Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 20080031
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Pain; Ponv; Fatigue
Keywords: laparoscopic cholecystectomy; pain; PONV; music; therapy; fatigue after elective laparoscopic cholecystectomy
MeSH Terms: conditions — Pain; Postoperative Nausea and Vomiting; Fatigue

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- music (Active Comparator)
  Interventions: Device: music pillow
- Pillow without music (Placebo Comparator)
  Interventions: Device: pillow without music

INTERVENTIONS:
Device: music pillow — according to randomisation patients will receive with/without music.
  Arms: music
Device: pillow without music — According to randomisation patients will receive a pillow with/without music
  Arms: Pillow without music

SUMMARY:
The study is undertaken to investigate whether relaxing music therapy before, during and after laparoscopic cholecystectomy has any effect on pain, PONV or fatigue and level of stress as measured by Cortisol and C reactive protein.

Patients will be scored according to those endpoints 1 and 3 hours after surgery and on day 1 and 7 post-OP.

ELIGIBILITY:
Inclusion Criteria:

* All patients going for laparoscopic cholecystectomy

Exclusion Criteria:

* Age below 18,
* Use of NSAID, morphine, steroids
* Disability
* Previous surgery in the past month
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2008-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Significant reduction in post operative VAS score | 1 week

SECONDARY OUTCOMES:
Significant reduction in Stress hormone level (Cortisol and C reactive protein) | 1 day

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - DaySurgical unit Regionshospital Randers, Randers
  - Regions Hospital Randers, Randers